CLINICAL TRIAL: NCT03323372
Title: Different Concentrations of Potassium Nitrate in In-office Tooth Bleaching Sensitivity: a Randomized Clinical Trial
Brief Title: Different Concentrations of Potassium Nitrate in In-office Tooth Bleaching Sensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Amazonas (Other)
Responsible Party: Principal Investigator, larissa alves de lima e souza, master student, Universidade Federal do Amazonas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UFAmazonas
Record Dates: First submitted 2017-10-02; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Tooth Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — potassium nitrate; Sodium Fluoride

STUDY DESIGN:
Intervention Model Description: The design of this randomized, double blind, intervention study was structured based on the CONSORT (Consolidated Standards of Reporting Trials) standards.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Active Comparator): In group 1 (G1-control), the operator applied a desensitizing gel based on 5% potassium nitrate and 2% sodium fluoride (Desensibilize KF 2% ®, FGM , Joinville, Santa Catarina, Brazil) with the aid of a custom silicone tray, which was made from a model obtained from the patient, with a vacuum plasticizer. A small layer of the gel was placed on the surface of the tray that was in contact with the vestibular face of the upper anterior teeth of the participants. The tray remained in position in the mouth for 10 minutes, according to the manufacturer's specifications.
  Interventions: Drug: 5% potassium nitrate and 2% sodium fluoride
- experimental group (Experimental): In group 2 (G2-intervention group), the operator applied a desensitizing gel containing 3% potassium nitrate and 0.25% sodium fluoride (Ultra EZ®, Ultradent Products Inc, South Jordan, UT, Estados Unidos) with the help of a tray in which the material is stored on the vestibular surfaces of the upper anterior teeth of the participants. The tray remained in position in the mouth for 15 minutes, according to the manufacturer's specifications.
  Interventions: Drug: 3% potassium nitrate and 0.25% sodium fluoride

INTERVENTIONS:
Drug: 3% potassium nitrate and 0.25% sodium fluoride
  Other Names: Ultra EZ
  Arms: experimental group
Drug: 5% potassium nitrate and 2% sodium fluoride
  Other Names: Desensibilize KF 2%
  Arms: control group

SUMMARY:
The aim of this randomized, double-blind controlled clinical study was to evaluate the absolute risk and intensity of sensitivity to dental bleaching in adults on the application of two different gels based on potassium nitrate and sodium fluoride from a prospective randomized clinical study.

DETAILED DESCRIPTION:
For this study, 56 volunteers who had an equal allocation rate between the groups (G1-control and G2-experimental) were selected for this study. Both gels act in the same way, the difference between them is the concentration. In both groups, the different desensitizing gels were applied to the vestibular surface of the anterior superior teeth with the aid of a tray, remaining in position according to the time specified by the manufacturers. In the control group, a gel based on 5% potassium nitrate and 2% sodium fluoride was used, while in the experimental group, the gel was based on 3% potassium nitrate and 0.25% sodium fluoride. After removal of the desensitizing gel, both groups were subjected to bleaching with 40% hydrogen peroxide gel for 40 minutes. Patients recorded an occurrence or not of dental sensitivity (SD) in a sensitivity diary for 48 hours. A Verbal Evaluation Scale (VRS) and a Visual Analogue Scale (VAS) were used for pain assessment. The values were organized into two categories: percentage of patients who presented SD at some time of treatment (absolute risk of sensitivity) and SD intensity. To evaluate the color before the first bleaching session, and after 7, 14 and 28 days, two methods were used: objective evaluation using the spectrophotometer and subjective evaluation using two color scales: Vita Classical and Vita Bleachedguide 3D-MASTER. An analysis of the data followed the intent-to-treat protocol and involved all randomly allocated participants. The absolute risk of SD was compared using Fisher's exact test (α = 5%). The Mann-Whitney test was used to compare the intensity of SD.

Student's t test was used to compare the color change. The level of significance adopted in all tests was 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older, of both sexes, who had to present at least six upper anterior teeth free of caries and restorations on the vestibular face, and at least one central or canine incisor showing coloration A2 or darker, evaluated in comparison to a visual value-oriented color scale of the teeth (Vita Classical®, Vita-Zahnfabrik- Germany).

Prior to the interventions, the signing of each participant's free and informed consent form (Appendix I) was obtained after due explanations about the nature of the study and the possible risks of the proposed treatments.

Exclusion Criteria:

* The individuals excluded from the study were: users of fixed orthodontic appliances, patients with periodontal disease, pregnant or lactating, with severe intrinsic stains on the teeth (spots on the use of tetracycline, fluorosis and depolluted teeth), consuming any Anti-inflammatory and anti-oxidant drugs, using desensitizing dentifrice and participants with previous history of SD or any associated pathology (bruxism, gingival recession, non-carious lesion with dentin exposure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-12-21; Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-20 (Actual)

PRIMARY OUTCOMES:
absolute risk of tooth sensibility | 28 days
  Patients recorded the occurrence or not of tooth sensitivity (TS) in a sensitivity diary. Participants were asked to register if they experienced DS during treatment and up to 48 hours after bleaching. The Analogic Visual Scale (AVS) was used to assess pain. Each item was scored 0-10 (0- no pain and 10- pain as bad as can be).

SECONDARY OUTCOMES:
sensitivity intensity | 28 days
  Patients were asked to record their perception of tooth sensitivity (TS) during the first and second bleaching sessions using the five-point Numeric Rating Scale (0 = none, 1 = mild, 2 = moderate, 3 = considerable, and 4 = severe]. Subjects were asked to record their experience with TS during the treatment, up to 1 h after bleaching, from 1 h to 24 h, and from 24 to 48 h after bleaching. They were also asked to record whether their experienced or not TS during the 30-day period after bleaching. As two bleaching sessions were performed, the highest score obtained in both bleaching sessions was considered for statistical purposes.
effectiveness of tooth whitening - objective | 28 days
  Color was recorded before the bleaching procedure, 7 days and 30 days after the end of the bleaching treatment using an objective method (Easyshade spectrophotometer, Vident, Brea, CA, USA). For each evaluation, three readings were performed using the CIELab system parameters, in which: L * indicates luminosity, a * represents color and saturation on the red-green axis and b * means color and saturation on the yellow-blue axis. Color evaluation was done in a room under artificial lightning conditions without interference from outside light. The color was checked at the middle third of the canine.
effectiveness of tooth whitening - subjective | 28 days
  Color was recorded before the bleaching procedure, 7 days and 30 days after the end of the bleaching treatment using a subjective (value-oriented shade guide Vita Classic). For subjective evaluation, the 16 color guides of the Vita Classical scale (Vita Zahnfabrik®, Bad Säckingen, Germany) were organized from the highest value (B1) to the lowest value (C4). Although the scale is not linear, it was organized by value representing a ranking for analysis purposes. Color evaluation was done in a room under artificial lightning conditions without interference from outside light. The color was checked at the middle third of the canine.

CONTACTS AND LOCATIONS:
Overall Officials: Leandro M Martins, doctorate, Study Chair — amazon federal university

IPD SHARING:
Plan to Share IPD: No